CLINICAL TRIAL: NCT01711450
Title: Randomised Double Blind Controlled Study of the Effectiveness of Paravertebral Nerve Block in Decreasing Analgesia Requirements and Improving Patient Experience During Interventional Hepatic Procedures.
Brief Title: Success of Paravertebral Blocks in Analgesia for Interventional Hepatic Procedures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Institutional Ethics Board concern regarding sham procedure, requiring modifications that are not feasible within the man-power limitations of our institution.
Sponsor: Richard Lindsay (Other)
Responsible Party: Sponsor-Investigator, Richard Lindsay, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Organization: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12-263-SDR
Record Dates: First submitted 2012-10-18; First posted 2012-10-22 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: Liver Neoplasms
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paravertebral block (Experimental): Paravertebral space will be needled and an anesthetic agent will be injected.
  Interventions: Procedure: Paravertebral block
- Control sham procedure (Placebo Comparator): Paravertebral space will be needled, but only normal saline injected.
  Interventions: Procedure: Control sham procedure

INTERVENTIONS:
Procedure: Paravertebral block — Injection of local anaesthesia into paravertebral space to provide analgesia
  Arms: Paravertebral block
Procedure: Control sham procedure — Injection of Normal saline into the paravertebral space
  Arms: Control sham procedure

SUMMARY:
This study is aimed at assessing whether performing a paravertebral block (a type of regional pain relief) can reduce the pain and anxiety patients experience during radiological procedures on the liver.

DETAILED DESCRIPTION:
Percutaneous procedures of the liver can be very painful and range from bliliary drain insertions to tumor ablation procedures. The study will randomize patients in two groups, one receiving a paravertebral nerve block prior to the procedure and one receiving a sham procedure in which saline will be injected in the paravertebral space. Pain scores and use of IV sedation will be monitored post procedure and both groups will be compared to assess whether paravetebral nerve blocks are effective at reducing pain in patients receiving such procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-pregnant female subjects, between the ages of 18 and 80 at the time of enrollment.

Subjects referred for liver/biliary interventions to the angiography department.

Written informed consent to participate in the study. Ability to comply with the requirements of the study procedures

Exclusion Criteria:

* Subjects who participated in an active stage of any drug, intervention or treatment trial within 30 days of enrollment.

Subjects with preexisting conditions, which, in the opinion of the investigator, interfere with the conduct of the study. Patients will only be excluded on this basis following discussion with another interventional radiologist.

Subjects who are uncooperative or cannot follow instructions. Mental state that may preclude completion of the study procedure or ability to obtain informed consent.

Pregnant or nursing female subjects. Patient who are to undergo liver biopsy or routine biliary tube exchange. Patients with neurological/spinal conditions, or a BMI over 40, that would prevent safe/effective or well-targeted paravertebral blockade.

Patient unable to tolerate the paravertebral block procedure, for example due to inability to lie prone

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-12; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Dose of intravenous sedation required during and after the procedure | 1 hour

SECONDARY OUTCOMES:
Improvement in analogue pain scoring after the procedure | 1 hour
Procedure duration | 1 hour
Complication rate of liver procedure | 24 hours
Complication rate of paravertebral block | 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lindsay, MB Bch, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Louis Boucher, MD, Study Director — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (2):
- Canada (2):
  - Royal Victoria Hospital, Montreal, Quebec
  - Montreal General Hospital, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No